CLINICAL TRIAL: NCT06194604
Title: Effectiveness of Instrument-Assısted Soft Tissue Mobılızatıon in Patients With Operated Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Levent Horoz, Asst Prof, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 118349
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Distal Radius Fractures; Instrument-assisted Soft Tissue Mobilization
Keywords: Instrument-assisted soft tissue mobilization; Distal Radius Fractures; edema; manuel therapy
MeSH Terms: conditions — Wrist Fractures; Edema

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and The outcomes assesor different persons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In addition to the routine physical therapy program, Instrument-assisted soft tissue mobilization will be applied 3 days a week, for a total of 18 sessions. Each session will last 5 minutes.
  Interventions: Device: Instrument-assisted soft tissue mobilization; Other: Routine rehabilitation programe
- Control group (Other): Only the routine physical therapy program will be applied.
  Interventions: Other: Routine rehabilitation programe

INTERVENTIONS:
Device: Instrument-assisted soft tissue mobilization — Instrumented soft tissue mobilization is a type of manual therapy method.Istrumented soft tissue mobilization aims to reduce fascial limitations by increasing circulation. Increases in localized blood flow and soft tissue realignment promote muscle function, increased normal joint movement, and decreased pain.
  Arms: experimental group
Other: Routine rehabilitation programe — Routine rehabilitation programe consisting of stretching and strengthening exercises will be applied.

SUMMARY:
Distal radius fractures are the most common fractures when looking at upper extremity fractures . The incidence of distal radius fractures is increasing day by day, and when looking at the databases of various countries, the annual prevalence reaches 70,000 in the UK and 640,000 in the USA. Most of them are related to osteoporosis, and if appropriate treatment is not given, they cause loss of work capacity, permanent disability, and limitation in daily activities . There are publications showing that short immobilization and appropriate rehabilitation after surgery provide good clinical results. In cases that are not properly rehabilitated after surgery, there may be an average delay of 12 weeks in returning to normal life and returning to work. When patients who were given early mobilization and rehabilitation after surgery were examined, it was observed that there was a significant improvement in wrist functions, range of motion, and grip strength . Instrumented soft tissue mobilization is a unique soft tissue mobilization combined with active mobility and stretching exercises that is prescribed to increase joint range of motion in patients with musculoskeletal injuries. The various sizes and beveled edges of the stainless steel instruments allow physical therapists to tailor the treatment to different muscle structures that experience myofascial restrictions. Instrumented soft tissue mobilization aims to reduce fascial limitations by increasing circulation. Increases in localized blood flow and soft tissue realignment promote muscle function, increased normal joint movement, and decreased pain.

DETAILED DESCRIPTION:
Instrument-assisted soft tissue mobilization (IATSM) has been studied in musculoskeletal system diseases of the upper extremity, lower extremity and spine. The first randomized controlled study examining the effect of the IASTM technique in trigger point treatment was conducted in 2014. A recent review reports that interest in the IASTM technique in musculoskeletal diseases has increased in recent years, but there is not enough evidence to support its use. It has been reported that randomized controlled studies have a high bias rate and are of low quality. In a recent article, IASTM was applied to cases with limited joint range of motion due to elbow fracture. Bhosale et al. They reported its effectiveness on pain, pain-related disability and joint range of motion .

Reducing pain and edema after Distal Radius fracture is an important part of postoperative rehabilitation. Various mobilization methods have been applied to this patient population in the postoperative period. There is no study in the literature evaluating the effectiveness of adding IASTM to the postoperative rehabilitation program in patients who underwent surgery for distal radius fractures.

This study aimed to evaluate the effect of adding IASTM to the postoperative rehabilitation program on pain, edema, joint range of motion and functionality in patients who underwent surgery due to distal radius fracture.

ELIGIBILITY:
Inclusion Criteria:

* Having volar plate applied due to distal radius fracture being over 18 years old
* No major postoperative complications (such as neurovascular injury, hematoma)

Exclusion Criteria:

* presence of polytrauma
* Surgical intervention other than volar plate
* History of previous limb-related surgery
* Hemiplegia in the involved limb
* Contracture in the involved limb

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Day 0
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale. Patients are asked to indicate their pain level, with 0 points being no pain, 5 points being moderate pain, and 10 points being unbearable pain. Increased scores indicate higher pain levels. Activity and rest VAS will be evaluated.
Visual analog scale | 4th week
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale. Patients are asked to indicate their pain level, with 0 points being no pain, 5 points being moderate pain, and 10 points being unbearable pain. Increased scores indicate higher pain levels. Activity and rest VAS will be evaluated.
Visual analog scale | 6th week
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale. Patients are asked to indicate their pain level, with 0 points being no pain, 5 points being moderate pain, and 10 points being unbearable pain. Increased scores indicate higher pain levels. Activity and rest VAS will be evaluated.
Wrist joint range of motion | Day 0
  Wrist joint range of motion: Measurement of wrist joint range of motion (ROM) with a goniometer is the most frequently used method in clinical practice that provides objective evaluation and error-free measurement. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Wrist joint range of motion | 4th week
  Wrist joint range of motion: Measurement of wrist joint range of motion (ROM) with a goniometer is the most frequently used method in clinical practice that provides objective evaluation and error-free measurement. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Wrist joint range of motion | 6th week
  Wrist joint range of motion: Measurement of wrist joint range of motion (ROM) with a goniometer is the most frequently used method in clinical practice that provides objective evaluation and error-free measurement. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Circumference (mm) | Day 0
  Environmental Measurement; Both hands and wrists of the patient will be measured with the help of a tape measure using the figure of eight method. The cm difference between both upper extremities will be recorded.
Circumference (mm) | 4th week
  Environmental Measurement; Both hands and wrists of the patient will be measured with the help of a tape measure using the figure of eight method. The cm difference between both upper extremities will be recorded.
Circumference (mm) | 6th week
  Environmental Measurement; Both hands and wrists of the patient will be measured with the help of a tape measure using the figure of eight method. The cm difference between both upper extremities will be recorded.

SECONDARY OUTCOMES:
Gross Grip Strength: | Day 0
  Jamar dynamometer wii use to evaluate gross grip strength.Higher values indicate increased grip strength
Gross Grip Strength: | 4th week
  Jamar dynamometer wii use to evaluate gross grip strength.Higher values indicate increased grip strength
Gross Grip Strength: | 6 th week
  Jamar dynamometer wii use to evaluate gross grip strength.Higher values indicate increased grip strength
Patient-Rated Wrist Evaluation (PRWE) questionnaire | Day 0
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire.High scores indicate functional impairment designed to measure wrist pain and disability in activities of daily living.The maximum score that can be obtained from the pain subscale is 50 and the minimum is 0.
  The maximum score that can be obtained from the function subscale is 50 and the minimum is 0.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 4th week
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire.High scores indicate functional impairment designed to measure wrist pain and disability in activities of daily living.The maximum score that can be obtained from the pain subscale is 50 and the minimum is 0.
  The maximum score that can be obtained from the function subscale is 50 and the minimum is 0.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 6 th week
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire.High scores indicate functional impairment designed to measure wrist pain and disability in activities of daily living.The maximum score that can be obtained from the pain subscale is 50 and the minimum is 0.
  The maximum score that can be obtained from the function subscale is 50 and the minimum is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Horoz, Asst Prof, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Research and Training Hospital, Kırşehir, Kişrsehşr, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No